CLINICAL TRIAL: NCT06091124
Title: A Prospective, Single-arm, Exploratory Study on the Efficacy and Safety of Neoadjuvant Adebrelimab Plus Etoposide and Cisplatin in Patients With Neuroendocrine Bladder Carcinoma
Brief Title: Neoadjuvant Adebrelimab Plus Etoposide and Cisplatin in Neuroendocrine Bladder Carcinoma
Acronym: NEOBLAST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2023-0177
Record Dates: First submitted 2023-10-14; First posted 2023-10-19 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Neuroendocrine Carcinoma of the Bladder; Bladder Cancer
Keywords: Neuroendocrine Carcinoma of the Bladder; Neoadjuvant Therapy; Adebrelimab; Etoposide; Cisplatin
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Etoposide; Cisplatin; Cystectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Adebrelimab Plus Etoposide and Cisplatin Followed by Radical Cystectomy (Experimental): The study population will include male and female patients over the age of 18 with invasive (cT1-cT4) neuroendocrine carcinoma of the bladder, with or without urothelial component (neuroendocrine component should be >50%). Patients with resectable N1-3 disease (judged by investigators) are eligible. Patients should be fit to undergo cystectomy with normal function of vital organs.
  Participants will be intravenously treated with adebrelimab (1200mg, day 1) in combination with etoposide (0.1g, day 1-3) and cisplatin (35mg/m2, day 1-2) every 21 days for a maximum of 4 cycles. Radical cystectomy, lymph node dissection and urine diversion will be performed after the completion of therapy.
  Interventions: Drug: Adebrelimab; Drug: Etoposide; Drug: Cisplatin; Procedure: Radical Cystectomy

INTERVENTIONS:
Drug: Adebrelimab — Adebrelimab 1200 mg IV on Day 1, once every 3 weeks for up to 4 cycles (each cycle = 21 days)
  Other Names: SHR-1316; HTI-1088
Drug: Etoposide — Etoposide 0.1g IV on Days 1-3, once every 3 weeks for up to 4 cycles (each cycle = 21 days)
  Other Names: VP-16; Vepesid; Toposar
Drug: Cisplatin — Cisplatin 35mg/m2 IV on Days 1-2, once every 3 weeks for up to 4 cycles (each cycle = 21 days)
  Other Names: Cis-Diaminedichloroplatinum; CDDP
Procedure: Radical Cystectomy — Radical cystectomy should be performed within 4-6 weeks after completion of last dose
  Other Names: RC

SUMMARY:
The goal of this clinical trial is to learn about the efficacy and safety of neoadjuvant adebrelimab plus etoposide and cisplatin in patients with neuroendocrine bladder carcinoma. The main questions it aims to answer are:

* The pathologic complete response rate at radical cystectomy
* Safety and tolerability of combination therapy Participants will be treated with a combination therapy of adebrelimab, etoposide, and cisplatin before radical cystectomy, with a maximum of 4 cycles.

DETAILED DESCRIPTION:
This is an prospective, single-arm, open-label clinical study of neoadjuvant adebrelimab in combination with etoposide and cisplatin in patients with neuroendocrine bladder carcinoma. Approximately 22 participants will be enrolled in this study to evaluate the efficacy and safety of neoadjuvant adebrelimab, cisplatin and etoposide.

The study population will include male and female patients over the age of 18 with invasive (cT1-cT4) neuroendocrine carcinoma of the bladder, with or without urothelial component (neuroendocrine component should be >50%). Patients with resectable N1-3 disease (judged by investigators) are eligible. Patients should be fit to undergo cystectomy with normal function of vital organs.

Participants will be intravenously treated with adebrelimab (1200mg, day 1) in combination with etoposide (0.1g, day 1-3) and cisplatin (35mg/m2, day 1-2) every 21 days for a maximum of 4 cycles. Radical cystectomy, lymph node dissection and urine diversion will be performed after the completion of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged ≥18 years and ≤75 years.
* ECOG performance status of 0 - 2.
* Histologically confirmed invasive neuroendocrine carcinoma with or without urothelial carcinoma, with a neuroendocrine carcinoma component of >50%; Formalin-fixed paraffin-embedded (FFPE) specimens (preferred) or at least 15 unstained, freshly cut, continuous slides should be submitted with related pathology reports prior to study enrollment. If fewer than 15 slides are available, patients may still be eligible for enrollment after confirmation by the principal investigator. If a tumor tissue section is not available, the tumor tissue must be obtained from the biopsy performed at the time of screening.
* Clinical stage T1-T4a N0 M0 (CT/MRI ± PET/CT) If the clinical stage is T1-4a N1-3 M0, it needs to be judged by the investigator. If cystectomy can still be performed, participants can be included in the study.
* Expected survival longer 3 months.
* Normal function of vital organs (14 days prior to enrollment). Meet the following criteria:

  1. Blood routine examination:

     HB≥90 g/L; ANC≥1.5×109 /L; PLT≥100×109 /L.
  2. No functional organic disease:

T-BIL≤1.5×ULN (upper limit of normal); ALT and AST≤2.5 x ULN; Serum creatinine ≤2×ULN, or endogenous creatinine clearance > 20 mL /min (Cockcroft-Gault formula); International Standardized ratio (INR), activated partial thromboplastin time (aPTT) : ≤1.5× ULN.

* Fertile males or females must use a highly effective contraceptive approach (such as oral contraceptives, intrauterine devices, abstinence or barrier contraception combined with spermicides) during the trial and continue contraception for 12 months after the end of treatment.
* Participants who voluntarily join the study, sign informed consent, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

* Prior anti-PD-1, anti-PD-L1 or anti-CTLA-4 therapy.
* Prior drug therapy for cancer, except:

Intravesical chemotherapy or immunotherapy ended at least 1 week before the start of study.

* Prior radiotherapy for bladder cancer.
* Participants allergic to adebrelimab and its components.
* Participants who have received other antitumor therapy or immunomodulatory therapy (including corticosteroid therapy, immunotherapy) or participated in other clinical studies within 4 weeks before the start of study treatment, or have not recovered from previous toxicity (except for 2 degree alopecia and 1 degree neurotoxicity).
* Pregnant or lactating females.
* HIV Positive.
* Participants with active hepatitis B or C:

For participants with HBsAg or HBcAb positive and detected HBV DNA copy number (quantitative detection limit is 500IU/ml, or reach the positive value of copy number detected by the research center), HBV DNA must be tested for screening in such patients.

Participants positive for HCV antibodies were enrolled in this study only if the PCR test for HCV RNA was negative.

* Active tuberculosis.
* Active autoimmune disease that requires systemic treatment within the past 2 years (such as disease-modulating drugs, corticosteroids, or immunosuppressive drugs). Replacement therapy (such as thyroxine, insulin, or physiologic corticosteroid replacement therapy for renal or pituitary insufficiency) are accepted.
* Other serious, uncontrolled medical conditions that may affect protocol adherence or interfere with interpretation of results. These include active opportunistic or progressive (severe) infections, uncontrolled diabetes, cardiovascular disease (heart failure as defined by the New York Heart Association scale as grade III or IV, cardiac conduction block above grade II, myocardial infarction within the last 6 months, unstable arrhythmia or unstable angina, cerebral infarction within the last 3 months, etc.), or pulmonary disease (interstitial pneumonia, Obstructive pulmonary disease and a history of symptomatic bronchospasm).
* Those who received live vaccine within 4 weeks prior to the start of treatment (seasonal influenza vaccines are usually inactivated and therefore permitted for use). Intranasal vaccines are live vaccines, so they are not allowed to be used).
* Prior allogeneic hematopoietic stem cell transplantation or solid organ transplantation.
* History of psychotropic substance abuse and cannot abstain or have a history of mental disorders.
* Pleural fluid or ascites associated with clinical symptoms or requiring symptomatic management.
* Participants with other malignancies that have not healed in the past 5 years, excluding apparently cured malignancies, or curable cancers such as basal or squamous cell skin cancer, localized low-risk prostate cancer, cervical carcinoma in situ, or breast carcinoma in situ.
* Concomitant upper tract urothelial carcinoma (pelvis and ureter urothelial carcinoma).
* Other severe, acute, or chronic medical or psychiatric disorders, or laboratory abnormalities that, in the investigator's opinion, may increase the risks associated with study participation or that may interfere with the interpretation of the study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (ypCR) at cystectomy | At the time of radical cystectomy (within 18 weeks of the first dose)
  The number of participants with pathologic complete responses (ypCR) at cystectomy. Pathologic complete response is defined as post-treatment stages of T0N0M0 .
Safety and tolerability of combination therapy and radical cystectomy | Up to 2 years
  The number of participants experiencing treatment-related adverse events, defined by NCI CTCAE 5.0

SECONDARY OUTCOMES:
Pathologic downstage at cystectomy | At the time of radical cystectomy (within 18 weeks of the first dose)
  The number of participants with pathological downstage at cystectomy. Pathologic downstage response is defined as downstaged T stage or N stage at cystectomy .
Progression Free Survival | Up to 2 years
  Defined by time from day of first treatment to disease progression
Cancer Specific Survival | Up to 2 years
  Defined by time from day of first treatment to death of the disease
Overall Survival | Up to 2 years
  Defined by time from day of first treatment to death

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi'an, Shaanxi
  - RenJi Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Chengdu, Sichuan
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No